CLINICAL TRIAL: NCT02953067
Title: A Multi-center, Prospective, Randomised Study of Treatment of Lisfranc Injuries
Brief Title: Study of Treatment of Lisfranc Injuries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to reach the required sample size
Sponsor: Tampere University Hospital (Other)
Collaborators: Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Heidi Haapasalo, MD, PhD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R11152
Record Dates: First submitted 2016-10-24; First posted 2016-11-02 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Foot Injury
MeSH Terms: conditions — Foot Injuries | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Open reduction and internal fixation (Active Comparator): After operative treatment non-weightbearing cast immobilisation for 6 weeks. Cast will be changed after 2 weeks. After the 6 weeks cast will be replaced with orthotics. Orthotics will remain for 4 weeks.
  Interventions: Procedure: Open reduction and internal fixation
- Primary Arthrodesis (Active Comparator): After operative treatment non-weightbearing cast immobilisation for 6 weeks. Cast will be changed after 2 weeks. After the 6 weeks cast will be replaced with orthotics. Orthotics will remain for 4 weeks.
  Interventions: Procedure: Primary arthrodesis
- Conservative treatment (Active Comparator): Non-weightbearing cast immobilisation for 6 weeks. Cast will be changed after 2 weeks. After the 6 weeks cast will be replaced with orthotics. Orthotics will remain for 4 weeks.
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Stratum 1: Conservative treatment versus open reduction and internal fixation Stratum 2: Open reduction and internal fixation versus arthrodesis
  Arms: Open reduction and internal fixation
Procedure: Primary arthrodesis — Primary arthrodesis versus ORIF
  Arms: Primary Arthrodesis
Procedure: Conservative treatment — Conservative treatment versus open reduction and internal fixation
  Arms: Conservative treatment

SUMMARY:
This trial is designed to compare different treatments on Lisfranc fractures. The trial consist of 2 different strata. Stratum 1: In mild injuries the comparison is between conservative treatment and operative treatment with open reduction and internal fixation (ORIF). Stratum 2: In severe injuries the comparison is between operative treatment with open reduction and internal fixation (ORIF) and primary arthrodesis. The primary outcome measure will be AOFAS Midfoot Score, and secondary outcome measure will be VAS Foot and Ankle.

DETAILED DESCRIPTION:
The aim of this study is to find out the most effective way to treat Lisfranc injuries

ELIGIBILITY:
Inclusion Criteria:

Stratum 1:

* Nondislocated fractures affecting tarsometatarsal (TMT) joints II and III
* Dislocation <5mm between medial cuneiforme and base of II metatarsal (MT)
* No fractures affecting TMT joints IV and V

Stratum 2:

* Affected joints TMT II- III + any other TMT
* Any dislocation >2mm (fracture or TMT joint)
* Dislocation >5mm between medial cuneiforme and base of II MT

Exclusion Criteria:

* Open fractures
* Extra-articular metatarsal (MT) fractures
* Extremely comminuted fractures with bone loss, and slight chance of gaining proper reduction with screws
* Patients with multiple fractures
* Patients with weak co-operation (dementia, alcohol use, etc.)
* Patients with significant neuropathy or some other neurological condition, diabetes and rheumatoid arthritis
* Patients with severe circulatory disorder of the lower limb
* Injuries over 14 days
* Patients with previous foot injury or surgery
* Pregnancy
* Patients who refuse to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
AOFAS Midfoot Scale | 12 months
  Between group difference in the functional outcome of the foot measured with AOFAS Midfoot Scale which is a subjective and objective evaluation of the midfoot based on questions in function (45 points), pain (40 points), and alignment (15 points) with a total score between 0 (worst score) and 100 (perfect score).
AOFAS Midfoot Scale | 24 months
  Between group difference in the functional outcome of the foot measured with AOFAS Midfoot Scale which is a subjective and objective evaluation of the midfoot based on questions in function (45 points), pain (40 points), and alignment (15 points) with a total score between 0 (worst score) and 100 (perfect score).

SECONDARY OUTCOMES:
VAS Foot and Ankle | 12 months
  Between group differences in pain and function of the foot measured with Visual Analog Scale of the Foot and Ankle (FA VAS). FA VAS scale is a self-administered patient questionnaire based on 20 questions in three different question categories (pain, function and other complaints). The total value of all questions is 2000. This total value is divided with 20 resulting in a possible score from 0 to 100 points, where 100 is the perfect score.
VAS Foot and Ankle | 24 months
  Between group differences in pain and function of the foot measured with Visual Analog Scale of the Foot and Ankle (FA VAS). FA VAS scale is a self-administered patient questionnaire based on 20 questions in three different question categories (pain, function and other complaints). The total value of all questions is 2000. This total value is divided with 20 resulting in a possible score from 0 to 100 points, where 100 is the perfect score.
VAS Pain | 6 weeks
  Between group difference in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).
VAS Pain | 10 weeks
  Between group differences in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).
VAS Pain | 4 months
  Between group differences in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).
VAS Pain | 6 months
  Between group differences in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).
VAS Pain | 12 months
  Between group differences in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).
VAS Pain | 24 months
  Between group differences in foot pain measured with Visual Analog Scale with a score of zero (no pain) to 100 (worst possible pain).

OTHER OUTCOMES:
Additional procedures or complications | up to 24months
  Number of patients with any additional procedure or complication of the treatment (implant removal, implant failure, any other reason of reoperation or complication of the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki-Jussi Laine, MD; PhD, Study Chair — Tampere University; Tiina Kaistila, MS, Study Chair — Tampere University; Ville Mattila, Professor, Study Chair — Tampere University; Antti Paakkala, MD;PhD, Study Chair — Tampere University; Heikki Mäenpää, Docent, Study Chair — Tampere University; Mikko Kirjavainen, MD; PhD, Study Chair — Dextra Fertility Clinic; Janne Jousmäki, MD, Study Chair — Seinajoki Central Hospital; Olli Väistö, MD; PhD, Study Chair — Seinajoki Central Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ponkilainen V, Maenpaa H, Laine HJ, Partio N, Vaisto O, Jousmaki J, Mattila VM, Haapasalo H. Open Reduction Internal Fixation vs Primary Arthrodesis for Displaced Lisfranc Injuries: A Multicenter Randomized Controlled Trial. Foot Ankle Int. 2024 Jun;45(6):612-620. doi: 10.1177/10711007241232667. Epub 2024 Mar 14. PMID 38482816
- [Derived] Ponkilainen VT, Mattila VM, Laine HJ, Paakkala A, Maenpaa HM, Haapasalo HH. Nonoperative, open reduction and internal fixation or primary arthrodesis in the treatment of Lisfranc injuries: a prospective, randomized, multicenter trial - study protocol. BMC Musculoskelet Disord. 2018 Aug 21;19(1):301. doi: 10.1186/s12891-018-2222-4. PMID 30126393